CLINICAL TRIAL: NCT04638387
Title: Nuclear Factor Erythroid 2-Related Factor 2 (Nrf2) Activation, Mobility, and Energetics: A Pilot and Feasibility Clinical Trial of PB125 Treatment for Improving Musculoskeletal and Pain Outcomes in Osteoarthritis
Brief Title: PB125, Osteoarthritis, Pain, Mobility, and Energetics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: pandemic limited recruitment; funding ran out
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Karyn Hamilton, Professor, Colorado State University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 19-9100H
Record Dates: First submitted 2020-11-12; First posted 2020-11-20 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee; Muscle Weakness; Pain, Joint
MeSH Terms: conditions — Osteoarthritis, Knee; Muscle Weakness; Arthralgia | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Primary comparisons will be between pre-test and post-test measures. We had initially planned control group comparisons as well, but the pandemic has cut this pilot study short of budget and time. Therefore, the primary comparisons will now be pre-test to post-test to maximize the number of participants enrolled to receive the experimental treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know if they are receiving PB125 or placebo. Participants will complete pain surveys. Team members making measurements of mobility and mitochondrial energetics will not know if participants or samples are PB125 or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB125 (Experimental): Twice daily oral administration of 1 capsule of PB125 (Pathways Bioscience). Treatment will last 12 weeks.
  Interventions: Dietary Supplement: PB125
- Placebo (Placebo Comparator): Twice daily oral administration of 1 capsule of rice flour placebo (Pathways Bioscience). Treatment will last 12 weeks. Because of pandemic restricting study time frame, enrollment will favor the experimental arm in this pilot study
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PB125 — Nrf2 activator containing active ingredients carnosol, withaferin A, and luteolin.
  Arms: PB125
Dietary Supplement: Placebo — Placebo comparator to P125
  Other Names: Flour
  Arms: Placebo

SUMMARY:
Nuclear factor erythroid 2-related factor 2 (Nrf2) is an important regulator in the body. It controls how well cells protect themselves against stress. PB125 (Pathways Bioscience) is a plant based activator of this important regulator Nrf2. PB125 is made up of three plant extracts (rosemary, ashwagandha, and Sophora japonica) so that it contains these things; 1. Carnosol, 2. Withaferin A, and 3. Luteolin. Carnosol comes from rosemary leaves. Rosemary is a spice often used in Italian foods and grown in many herb gardens all around Fort Collins. Withaferin A comes from the medicinal plant Withania somnifera, also called ashwagandha. Ashwaganda is commonly known as "Indian Winter cherry" or "Indian Ginseng" and it is one of the most important herbs of Ayurveda (the traditional system of medicine in India) used for millennia. Finally, luteolin is found widely in plants including those present in the diet (peppers, onions, celery, herbs/spices). Some people purchase these herbs commercially, and take them on their own for a variety of purposes. Typically, when you buy them, they will be in much higher doses than they are in PB125. What makes PB125 different is that very low doses of each of the 3 components work together-synergistically-to activate Nrf2 and increase the ability of cells to respond to stress. It is unknown if there are any benefits to taking PB125 and the risks are currently unknown. The purpose of this study is to examine changes in muscle, in joint pain, in mobility (standing and walking) and in leg strength that occur after consuming PB125 every day for 3 months. We want to make these measurements in people who have been diagnosed with mild to moderate osteoarthritis-a degenerative joint disease-in their knees.

DETAILED DESCRIPTION:
Preventing or slowing age-related decline in musculoskeletal function is important for maintaining mobility and independence. In the US, osteoarthritis (OA) is the primary cause of disability in adults, with no medical or surgical therapeutic intervention known to restore the degenerated cartilage. The loss of skeletal muscle mass and function with age, is also linked to increased risk of other diseases, risk of falls, and decreased quality of life. Therefore, OA and muscle loss together are primary contributors to age-related decreases in mobility and independence. Evidence suggests a decrease in muscle quality is associated with or precedes primary knee OA, suggesting that these two conditions may share a common cause. We will treat 50-65 year old people with mild or moderate OA in both knees, and reported loss of muscle strength, with a supplement already available for use in humans to reduce oxidative stress and inflammation. The supplement is called PB125. In this pilot clinical trial, we will measure the ability of muscle to make energy, measure mobility (walking and standing) and strength, and assess pain following PB125 or placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* bilateral knee osteoarthritis

Exclusion Criteria:

* smoking
* pregnant/breastfeeding
* BMI >30
* known liver, renal, heart disease, diabetes, autoimmune disease, cancer
* use of methotrexate, etanercept, infliximab, leflunomide, plaquenil
* recent serious illness
* intraarticular stem cell injection
* intraarticular steroid or hyaluronic acid injection within 4 months
* current enrollment in another trial of investigational drugs
* known hypersensitivity to ashwagandha, luteolin, rosemary, or rice flour
* use of anticoagulants or known bleeding disorder
* unwillingness to comply with protocol
* plans for knee replacement in the next 3 years
* unable to complete mobility testing without ambulatory aid
* unable to climb 1-2 flights or stairs without stopping/shortness of breath/discomfort
* blood product transfusion within 30 days
* unable to provide legal consent

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Mobility-6 min self-paced walk | Change from baseline at 12 weeks
  Change in Distance walked
Mobility-sit to stand | Change from baseline at 12 weeks
  Change in Time for 5 sit to stand repetitions
Mobility-static balance | Change from baseline at 12 weeks
  Yes/No ability to complete 30 sec trials with eyes open or closed on firm and foam surfaces
Mobility-6 min fast-paced walk | Change from baseline at 12 weeks
  Change in Distance walked
Intermittent and Constant Knee Pain | Change weekly for 12 weeks
  Weekly change in Intermittent and Constant Pain Score (ICOAP) 11 question survey of pain on a 0-4 scale
Energetics-Submaximal Oxygen Consumption | Change from baseline at 12 weeks
  Change in oxygen (O2) flux in permeabilized muscle fibers at submaximal adenosine diphosphate (ADP) concentrations
Energetics-Maximal Oxygen Consumption | Change from baseline at 12 weeks
  Change in O2 flux in permeabilized muscle fibers at maximal ADP concentrations

SECONDARY OUTCOMES:
Energetics-hydrogen peroxide emission | Change from baseline at 12 weeks
  Change in Hydrogen peroxide emission in permeabilized muscle fibers
Bone Mineral Density | Change from baseline at 12 weeks
  Bone mineral density via dual x-ray absorptiometry (DEXA)
Knee Range of Motion | Change from baseline at 12 weeks
  Change in active and passive bilateral knee range of motion
Leg extensor strength | Change from baseline at 12 weeks
  Change in maximal force generated during knee extension

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

REFERENCES:
- See also: Study Flyer on Colorado State University Center for Healthy Aging Website — https://www.research.colostate.edu/wp-content/uploads/2020/07/Knee-Osteoarthritis-Study-in-Health-and-Exercise-Science.pdf